CLINICAL TRIAL: NCT02935335
Title: Relationship Between antimüllerian Hormone Measured by a Fully Automated Assay and the Initial Dose of HP-hMG (Menopur®) Prescribed for Infertile Women Undergoing Their First IVF/ICSI Cycle.
Brief Title: A Study to Measure Relationship Between Antimüllerian Hormone and Initial Dose of Menopur®
Acronym: AME
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000237
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Menopur® HP-hMG: Treatment according to routine clinical practice.
  Interventions: Drug: Menotrophin

INTERVENTIONS:
Drug: Menotrophin
  Other Names: Menopur® HP-hMG

SUMMARY:
AME is a non-interventional, prospective, longitudinal and multicenter study. This study aims to measure the relationship between antimüllerian hormone serum level (AMH), as measured by a fully automated assay and the initial dose of Menopur® HP-hMG 600 IU/mL prescribed for infertile women undergoing their first IVF/ICSI cycle in the current practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between [18-42] years.
* Both ovaries present.
* Regular menstrual cycles presumed to be ovulatory.
* Primary or secondary infertility of any origin for more than 12 months.
* Patient with at least one result of antimüllerian hormone (AMH) measured by a fully automated assay available before inclusion, and performed in the past 12 months before inclusion.
* Candidates eligible to a first IVF/ICSI cycle and for whom Menopur® HP-hMG 600 IU/mL has been prescribed.
* Having received oral and written information on the study, without any objections for the use of his/her anonymized data, and having signed a written Informed Consent Form.

Exclusion Criteria:

* Major uterine or ovarian morphological abnormalities or past ovarian surgery.
* Endometriosis stage III/IV.
* Polycystic ovarian syndrome.
* Major endocrine or metabolic abnormalities without treatment.
* Patient included in an interventional study assessing treatment for infertility.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Specialized fertility centers.
Sampling Method: Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Spearman correlation coefficient between Menopur® 600 IU/mL dose and AMH serum levels | At baseline (inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Hospital FOCH (there may be other sites in this country), Suresnes, France